CLINICAL TRIAL: NCT03674164
Title: Fertility Preservation With Ovarian Tissue Freezing
Acronym: PTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Julio Saumet-Chilito, Physician, Director of fertility preservation department, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 217-1341
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Cancer; Hematologic Disorder; Infertility; Ovarian Failure
MeSH Terms: conditions — Neoplasms; Hematologic Diseases; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ovarian Cryopreservation — Surgical ovarian removal and vitrification

SUMMARY:
The purpose of this study is to obtain ovarian tissue from female patients undergoing gonadotoxic treatments or gonadal ablating surgery, and that in consequence may see their future fertility impaired. Participants will be offered to preserve (freeze) and use ovarian tissue for the purpose of conceiving in the future.

Although, 86 live births have been reported with ovarian tissue cryo-preservation and grafting, the procedure is still considered experimental.

This research, will help us to learn and validate how to perform ovarian tissue cryo-preservation and thawing in the fertility preservation context.

DETAILED DESCRIPTION:
his Study will conducted at the Centre Hospitalier Universitaire Ste-Justine Collected ovarian tissue will only be for the patients own use.

Subjects will undergo surgical removal of their ovarian tissue, and the following categories will be invited to participate:

1. Patients have elected to have one or both ovaries removed for the treatment or prevention of disease.
2. Patients who have elected to have surgery to remove all or part of one or both ovaries for medical reasons where cryopreservation of the remaining limited portions of normal ovarian cortex is the only option for fertility preservation at the time (except that ovarian cortex from the ovary that contains the mass will not be cryopreserved).
3. Participants who have elected to have one or part of one ovary removed, solely for the purpose of fertility preservation because they are not candies to use standard fertility preservation technologies.

If the subject chooses to participate and consent, she will be assessed to determine her eligibility The subject will also have a serum AMH drawn for the evaluation of the ovarian reserve, and also infectious disease testing will also be performed per Health Canada guidelines.

The oophorectomie will be performed laparoscopically under general anesthesia. In patients' in whom it is medically unsafe or not feasible to complete the surgery laparoscopically, the patient and/or legal gardian may opt to proceed with a mini-laparotomy or laparotomy approach or may opt to stop the procedure and withdraw from the study at that time. This decision will be discussed with the patient and legal gardian during the consenting process and documented prior to the surgery. The procedural risk and treatment delays will be discussed with the primary treatment team in order to provide a better evaluation of the patients wellbeing. This procedure is performed for fertility preservation purposes only, but can potentially be coordinated with another procedure such as placement of a central line for future chemotherapy. In the event the subject is undergoing a surgical intervention for other indications, the oophorectomies could be coordinated at the same time.

A tissu sample will be evaluated by pathology for routine histologic evaluation. If the pathologist finds evidence of neoplasia in the ovarian tissue sample. All the tissue could be send to pathology for a more detailed examination. In this case, there will be no tissue available for the subject to use for fertility preservation.

Cryopreservation :

Ovarian tissue preparation:

1. Ovarian tissue will be transported from the operating room at the CHU Sainte-Justine to the Embryology laboratory at the REI department in a modified HTF supplemented with 10% supplement serum substitute (9922 SSS; Irvine Scientifc, Santa Ana, CA, USA) and deposed in a heated trait at 37 °C.
2. The ovarian cortex will be separated from the medulla and cut in tissue bands (0.5-1 x 0.5- 1cm, 1-2 mm)
3. Tissue washing with TCM 199 (Life technologies, Foster City, CA, USA) supplemented with 20% (v/v) SSS (milieu WS) and then exposed to three different vitrification solutions at room temperature.

Vitrification:

1. Ovarian tissue equilibration in TCM199 avec 10% (v/v) ethylene glycol (EG, Wako Pure Chemical Industries, Tokyo, Japan) et 20% (v/v) SSS for 5 minutes.
2. Ovarian tissue equilibration in TCM199 with 20%(v/v) EG and 20% (v/v) SSS for 5 minutes.
3. Ovarian tissue equilibration in TCM199 avec 35%(v/v) EG, 5% (w/v) polyvinylpyrrolidone (sigma-Aldrich, St. Louis, MO, USA) et 0.5 mol/l sucrose (Wako Pure Chemical industries) for 5 minutes.
4. Ovarian tissue bands will be installed on" Cryosupport " (BD Bioscience, San Jose, CA, USA) before immersion in liquid nitrogen.
5. Ovarian tissue bands will be stored in a cryo vial at -196°C.

The ovarian tissue bio-bank is located at the embryology laboratory in the REI department at the CHU Ste-Justine

Infectious disease screening:

As per Health Canada guidelines, patients will be screened for (VIH, VDRL, HBsAg, anti Hepatitis C, HTLV).

Study and safety data collection:

Adverse events after an elective oophorectomy will be identified according to the Health Canada criteria (www.hc-sc.gc.ca/ahc-asc/media/advisories-avis/reaction-eng.php#Drugs).

Data Collection :

1. Date of fertility preservation

   1. Intervention type
   2. Age
   3. Age at diagnosis
   4. Age at menarche
2. Diagnosis
3. Outcome: remission, relapse, or death
4. Gynaecological history
5. Obstetrical and neonatal outcomes
6. Treatment regimen associated with high risk of sterility
7. Choices regarding use of cryopreserved stored tissue for fertility restoration Fertility preservation outcome

Risks:

The potential risks of laparoscopy, laparotomy, and oophorectomy include injury to bowel, bladder, and blood vessels with need for subsequent repair. The chance of the subject requiring hospitalization for complication(s) is about 1%. In addition to the surgical risk, there are also inherent risks of general anesthesia. The subject's chance of dying from anesthesia is less than 1 in 10,000. The risk of injury with laparotomy is moderate. The subject, legal guardian, and/or parent(s) will be asked to sign the standard consent form for laparoscopy, and/or laparotomy and oophorectomy after the risks and benefits have been discussed. The subject, legal guardian(s), and/or parent(s) will also be asked by the anesthesiology team to sign an anesthesia consent form after risks and benefits have been discussed.

There is a risk that the ovary to be cryopreserved may be affected by cancer, disqualifying the subject from ovarian tissue freezing. Although care will be taken, damage to the removed ovarian tissue may occur during any part of the cryopreservation, shipping or storage process. The effects of cryopreservation and long term storage on human ovarian tissues are not known and possible damage to the tissues may occur; in this instance a future pregnancy may not occur. The birth defect(s) and/or genetic damage to any child who may be born following ovarian tissue cryopreservation procedure are also unknown. However, thousands of children have been born worldwide from frozen embryos and eggs and there has been no report of increased risk of birth defects in these children.

Benefits:

The patient participation in the study protocol may provide her with a means to restore her fertility and reproductive hormonal function. However, However, there is a significant possibility that there may be no direct benefit due to no utilization of the ovarian tissue, or that the ovarian tissue may not result in any live brith.

Costs: All expenses related to this procedure will be covered by the "Régie s'Assurance du Québec". Tissue storage is also covered for a period of five years.

ELIGIBILITY:
Inclusion Criteria:

1. Females, > 2 month and < 18 years of age
2. Undergo surgery, chemotherapy, drug treatment, and/or radiation for the treatment or prevention of a medical condition or malignancy expected to result in permanent and complete loss of subsequent ovarian function.
3. Or, have a medical condition or malignancy that requires removal of all or part of one or both ovaries.
4. Subject may have newly diagnosed or recurrent disease.
5. Subject who already has stored cryopreserved ovarian tissue in a frozen state prior to undergoing cancer treatments (surgery, chemotherapy or radiation) will be eligible for enrolment with informed consent.
6. Subject not eligible to standard fertility preservation
7. The subject and/or the subject's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies.

Exclusion Criteria:

1. Women with psychological, psychiatric or other conditions which prevent giving fully informed consent.
2. Women whose underlying medical condition significantly increases their risk of complications from anesthesia and surgery.
3. Women to whom the research intervention may decrease the survival or the treatment response to the underlying disease.
4. AMH (Anti Müllerian Hormone) <0.016 ng/dl
5. Women whose surgery is preformed outside the CHU Ste-Justine
6. Patients eligible to a standard fertility preservation procedure.

   -

Ages: 2 Months to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2019-09-10 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cryopreservation of ovarian tissu by vitrification | 5 years
  Measure the fertility rate of cryopreservation and grafting by ovarian tissue vitrification.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Saumet Chilito, MD, Principal Investigator — Physician
Locations (1):
- CHU Ste-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No